CLINICAL TRIAL: NCT00089310
Title: Intraoperative Sentinel Node Mapping In Non-Small Cell Lung Cancer
Brief Title: Sentinel Lymph Node Mapping in Detecting Cancer That Has Spread to Lymph Nodes in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CALGB-140203; U10CA031946 (NIH); CALGB-140203; CDR0000378197 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Technetium-99

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sentinal node mapping (Experimental)
  Interventions: Radiation: technetium-99

INTERVENTIONS:
Radiation: technetium-99 — 0.25 mCi in 4 equal doses

SUMMARY:
RATIONALE: Diagnostic procedures such as sentinel lymph node mapping may improve the ability to detect cancer that has spread to the lymph nodes.

PURPOSE: This clinical trial is studying how well sentinel lymph node mapping works in detecting cancer that has spread to the lymph nodes in patients who are undergoing surgery for stage I non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility and accuracy of intraoperative sentinel lymph node mapping using technetium Tc 99 sulfur colloid in patients with stage I non-small cell lung cancer.
* Determine the percentage of patients in which at least 1 positive sentinel lymph node is identified using this procedure.
* Determine the percentage of patients undergoing this procedure who are found to have positive sentinel lymph nodes with no metastases in other intrathoracic lymph nodes.

Secondary

* Determine the percentage of patients undergoing this procedure whose disease stage is upgraded due to detection of micrometastases in sentinel lymph nodes.
* Correlate the presence of micrometastases in sentinel lymph nodes with survival in patients undergoing this procedure.
* Determine the percentage of patients undergoing this procedure with "skip metastases" pattern (NZ) sentinel lymph nodes.

OUTLINE: This is a multicenter study.

Patients receive an intraoperative intratumoral injection of technetium Tc 99 sulfur colloid. At least 10 minutes later, patients undergo sentinel lymph node mapping using a gamma probe. Patients then undergo sentinel lymph node dissection and tumor resection. Pathology assays are performed using sentinel lymph node tissue, including hematoxylin and eosin staining, serial sections, and immunohistochemistry using the AE1/AE3/PCK2b cytokeratin antibody.

Patients are followed every 6 months for 2 years and then annually thereafter.

ELIGIBILITY:
1. Patients with clinical stage I lung cancer for whom surgical resection is planned are eligible. Histologic confirmation of lung cancer is not required prior to registration or surgical exploration. Preoperative mediatinoscopy is allowed but not required in those patients with indications for mediatinoscopy. It is preferred that that mediatinoscopy be done at a different setting (prior to registration), but the procedure may be done at the same setting as the lobectomy.
2. No prior therapy for this diagnosis.
3. No prior treatment with mediastinal radiation therapy.
4. Age ≥ 18 years of age.
5. ECOG performance status: 0-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-09; Primary Completion 2007-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Sentinel node identification | at time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D'Amico, MD, Study Chair — Duke University
Locations (12):
- United States (12):
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio

REFERENCES:
- [Result] Liptay MJ, D'amico TA, Nwogu C, Demmy TL, Wang XF, Gu L, Litle VR, Swanson SJ, Kohman LJ; Thoracic Surgery Subcommittee of the Cancer and Leukemia Group B. Intraoperative sentinel node mapping with technitium-99 in lung cancer: results of CALGB 140203 multicenter phase II trial. J Thorac Oncol. 2009 Feb;4(2):198-202. doi: 10.1097/JTO.0b013e318194a2c3. PMID 19179896